CLINICAL TRIAL: NCT01360307
Title: Psychometric Validation of the Spanish Version of the CUDOS Scale (Clinically Useful Depression Outcome Scale) in Major Depressive Disorder
Brief Title: Validation of the Spanish Version of the Clinically Useful Depression Outcome Scale (CUDOS) Scale
Acronym: CUDOS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NES-XXX-2011/1
Record Dates: First submitted 2011-05-16; First posted 2011-05-25 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Unipolar Depression
Keywords: psychometric validation; major depressive disorder; patient-reported outcome
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Major Depressive Disorder Patients

SUMMARY:
The Clinically Useful Depression Outcome Scale (CUDOS) is a brief, self-administered instrument that not only evaluates depressive symptoms but also both functioning and quality of life. The assessment of patients´ perspective may provide valuable information that could be lost if relaying only on clinician evaluation. The purpose of this study is to achieve a psychometric validation into Spanish of the CUDOS scale in patients with major depression disorder in a primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* Major depression disorder diagnosis according to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) criteria in the last 3 months
* Major depression disorder diagnosis according to Prime-MD criteria in the last 3 months

Exclusion Criteria:

* Be unable to understand and comply with the study requirements as judged by the investigator
* Participation in another trial prior to enrolment into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Clinically Useful Depression Outcome Scale | up to 12 weeks after a diagnoses of a major depressive disorder
  To analyze feasibility and reliability (internal consistency - Cronbach´s alpha) of the Spanish version of the scale

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale | up to 12 weeks after a diagnoses of a major depressive disorder
  To analyze convergent validity of the Spanish version of the CUDOS scale
SF 36 | up to 12 weeks after a diagnoses of a major depressive disorder
  To analyze correlation in quality of life -item 18 of the CUDOS scale
Patient Global Impression Scale | up to 12 weeks after a diagnoses of a major depressive disorder
  To analyze criterion validity of the Spanish version of the CUDOS scale
Social Occupational Functioning Scale | up to 12 weeks after a diagnoses of a major depressive disorder
  To analyze correlation in functioning -item 17 of the CUDOS scale
Clinically Global Impression Scale | up to 12 weeks after a diagnoses of a major depressive disorder
  To analyze criterion validity of the Spanish version of the CUDOS scale

CONTACTS AND LOCATIONS:
Locations (17):
- Spain (17):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Cadiz
  - Research Site, Córdoba
  - Research Site, El Vendrell
  - Research Site, Granada
  - Research Site, Huelva
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Nigrán
  - Research Site, Palma Mallorca
  - Research Site, Salamanca
  - Research Site, Terrassa
  - Research Site, Tudela
  - Research Site, Vigo